CLINICAL TRIAL: NCT03543397
Title: Relevance of Mammary MRI in the Preoperative Assessment of Ductal Carcinoma in Situ (DCIS)
Brief Title: MRI in Ductal Carcinoma in Situ (DCIS)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7013
Record Dates: First submitted 2018-02-26; First posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-02

CONDITIONS: Ductal Carcinomas
Keywords: ductal carcinomas; ductal carcinoma in situ (DCIS); MRI
MeSH Terms: conditions — Carcinoma, Ductal; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Compare the estimate of the lesional size in MRI to that in mammography, taking as a reference the definitive anatomo-pathological size

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 ans
* Woman with DCIS

Exclusion Criteria:

* Age ≥18 ans)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Woman with DCIS
Sampling Method: Non-Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2018-02-26 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
The investigators compare the estimate of the lesional size in MRI to that in mammography, taking as a reference the definitive anatomo-pathological size | The period from January 1st, 2017 to December 31st, 2017 will be examined]
  Patients hospitalized at Strasbourg University Hospital in 2017

CONTACTS AND LOCATIONS:
Overall Officials: Marie Noëlle ROEDLICH, MD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service de Radiologie 1, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No